CLINICAL TRIAL: NCT02157103
Title: A Phase II Study of Subcutaneous Bevacizumab in Relapsed / Progressive Glioblastoma
Brief Title: A Study of Subcutaneous Bevacizumab in Relapsed / Progressive Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Read, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00062998; Winship2299-12 (Other: Winship Cancer Institute)
Record Dates: First submitted 2014-02-14; First posted 2014-06-05 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Glioblastoma
Keywords: GBM; Glioblastoma; Bevacizumab; Avastin; Subcutaneous
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Cycle 1 (each cycle is 3 weeks): Bevacizumab 25 mg in 1 ml subcutaneously daily.
  Interventions: Drug: Bevacizumab 25 mg in 1 ml subcutaneously daily

INTERVENTIONS:
Drug: Bevacizumab 25 mg in 1 ml subcutaneously daily — Bevacizumab delivered by subcutaneous injection instead of intravenous infusion.
  Other Names: Avastin

SUMMARY:
STUDY BACKGROUND:

This research will involve patients with glioblastoma. The drug bevacizumab (Avastin) is FDA approved for the treatment of glioblastoma that gets worse after standard therapy. For glioblastoma, bevacizumab is given by vein every 14 days. The purpose of this study is to see if bevacizumab works as well when it is given as a daily subcutaneous shot as it does when given intravenously. A subcutaneous shot is like an insulin shot or a heparin shot. The dose of bevacizumab given on this study is in total slightly lower than the FDA approved dose for glioblastoma.

STUDY DESCRIPTION:

About 10 people will take part in the study. Participants or caregivers will be educated on injection and given prefilled syringes to take home. Participants or caregivers will administer bevacizumab subcutaneously each day. The bevacizumab will be stored in the refrigerator.

Follow up visits will be weekly for the first 3 weeks, then every 3 weeks. After 18 weeks, the follow up interval can be increased to every 6 weeks at the treating physician's discretion.

Participants can keep taking the bevacizumab until:

* Tests show that they are not benefiting from it,
* The participant has a bad side effect related to study treatment,
* The participant can no longer comply with study requirements, or
* The participant or doctor feels it is no longer in the participant's best interest.

DETAILED DESCRIPTION:
1.1 Primary Aim: To describe MRI response rate as regards edema and enhancement of glioblastoma and radiation- related brain enhancement when treated with subcutaneous (SQ) bevacizumab daily. See section 11 for detail on response assessment.

1.2 Secondary Aims: 1.2.1 To characterize toxicities of SQ bevacizumab. 1.2.2 To describe response rate as per primary aim (above) in study participants who discontinue SQ bevacizumab for any reason and go on to receive treatment with standard IV bevacizumab or bevacizumab-containing combination.

2 BACKGROUND 2.1 Bevacizumab is a monoclonal antibody cancer therapeutic which targets vascular endothelial growth factor (VEGF) and which has been FDA approved for the treatment of glioblastoma. Clinical trials of bevacizumab in glioblastoma multiforme (GBM) patients documented edema and enhancement response rates between 75 and 100%, with consequent improvement in neurologic symptoms and decrease in corticosteroid requirements.(1-3) The FDA approval was based on response rate; there has not been proof that bevacizumab prolongs survival in GBM patients. The related VEGF antagonist cediranib can decrease brain edema in a manner comparable to bevacizumab(4) but failed to prolong survival in GBM patients in a recent phase III study.(5) Thus bevacizumab remains strictly palliative for GBM patients, a disease which in any case is not thought to be curable with available treatments.

2.2 Most monoclonal antibody therapeutics remain effective when given subcutaneously instead of intravenously.(6-9) Preclinical animal data show this to be true for bevacizumab as well, with 100% bioavailability for SQ as compared to IV administration.(10) In a mouse tumor model, SQ bevacizumab produced better antitumor effects than intravenous bevacizumab.(11) Some treatments are also less toxic when given subcutaneously - a recent example is bortezomib, which produces less neuropathy when given SQ instead of IV but is just as effective against myeloma.(12) This is presumably because of lower peak doses. There is no published correlation between dose of bevacizumab and incidence of the common side effects, which include hypertension and proteinuria, as well as less common but more dangerous toxicities such as gut perforation. If these toxicities relate to peak doses obtained after IV administration, it may be that they are less frequent in a dosing scheme in which SQ administration yields a low sustained and stable dose. It is not clear what SQ dose of bevacizumab is necessary to obtain benefit in GBM. Although the FDA approved dose is 10mg/kg every 14 days, earlier European GBM studies used 5mg/kg every 14 days and produced similar response rates.(1) This uncertainty about the required dose is, in fact, true for all the diseases in which bevacizumab is used; an example can be seen in two simultaneously published phase III ovarian cancer studies, one of which used bevacizumab maintenance at 15mg/kg every 3 weeks and the other half that dose at 7.5mg/kg every 3 weeks, with the lower dose study actually obtaining improved survival for participants as compared to the higher.(13, 14) It is possible that at least in GBM, lower doses might be better. Some theorize that the hypoxia produced by antiangiogenic treatments promote a more aggressive, infiltrative tumor phenotype. There is some thought that a less complete blockade of VEGF would decrease consequent hypoxia and conversion to this aggressive phenotype.(15) A recent retrospective series reported that GBM patients who encounter bevacizumab toxicity and undergo dose reduction have longer survival than contemporaneously treated GBM patients who continue at 10mg/kg every 14 days.(16) Thus it is ethical and perhaps even beneficial to explore lower doses of bevacizumab in the treatment of GBM.

2.3 The rapid and nearly universal response rate in GBM patients as regards enhancement and edema together with the direct palliative benefit of bevacizumab monotherapy makes this an excellent population to study an alternate dosing scheme. In this study the investigators propose to study subcutaneous bevacizumab for the treatment of patients with GBM and progressive edema representing tumor progression or symptomatic radiation aftereffects. All participants will receive the same dose of 25 mg SQ daily, which would translate into 350 mg over 14 days or 5mg/kg/14 days for a 70 kg patient - the same total dose used in the European GBM series and the same dose as is used to treat metastatic colon cancer. Bevacizumab solution is known to be stable in refrigerated prefilled syringes(17), and participants would take these home, injecting themselves after the manner of low molecular weight heparin. Participants would receive weekly toxicity assessment, and MRI at 3 weeks looking for evidence of response in terms of reduction of enhancement and edema; see section 11. Those participants with response would continue on SQ bevacizumab as long as they continued to experience clinical benefit. Participants not responding, progressing after initial response or encountering toxicity specific to the subcutaneous route of injection or discontinuing study participation for any reason would be offered conversion to standard IV bevacizumab as standard of care or other treatments as appropriate and available. Improvement in enhancement / edema among participants converting to standard IV bevacizumab or bevacizumab containing combinations will be followed as a secondary endpoint.

2.4 The study would be done as a Simon 2 stage, with an expected response rate as regards enhancement / edema of 90%. If fewer than 5 of an initial 6 participants show response the study will end and the SQ route will be deemed ineffective. If >4 of 6 respond, then accrual will expand to a total of 13 patients. See section 10.1, below.

2.5 The convenience of a SQ regimen would benefit some patients with GBM. The current requirement for IV therapy requires the patient to travel to an oncology infusion center and have IV access placed every other week, which is arduous and cumbersome. In addition, if bevacizumab were effective SQ for patients with GBM, this would offer the prospect of SQ bevacizumab being studied in other diseases with the goal of devising all-outpatient regimens and liberating patients from the infusion center. Examples include ovarian cancer (for which maintenance bevacizumab monotherapy improves survival), hereditary hemorrhagic telangiectasia, and in combination with other subcutaneous or oral medicines (e.g. capecitabine, interferon) for the treatment of metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Participants with glioblastoma are eligible for this study. These will include

  * Those with a histologically proven diagnosis of glioblastoma who have developed new changes on MRI following primary treatment.
  * Those who received primary treatment for a histologically proven lower grade (2 or 3) glioma and who now progress with radiographic characteristics of transformed glioma.
* Disease status: Patients must have abnormal enhancement on contrast enhanced MRI of the brain. They must be patients for whom bevacizumab is indicated and appropriate, as drug will be charged to insurance.

  * Participants with newly detected enhancement are eligible, with bevacizumab treatment hoped to prevent symptoms.
  * Participants with stable enhancement / edema are eligible if they require corticosteroids to control symptoms, and it is thought bevacizumab treatment might allow lowering of the corticosteroid dose or improvement of symptoms.
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-3.
* Age: Greater than 18 years.
* Life expectancy: > 3 months.
* Prior therapy:

  * Anti-VEGF treatments: 3 months must have elapsed between any prior anti-VEGF treatment (for example, given as a component of primary treatment) and study participation. These therapies include bevacizumab, cediranib, axitinib, sunitinib as well as other therapeutics targeting VEGF.
  * Other anti-cancer treatments: Treatments in this category include chemotherapy and targeted therapies not targeting VEGF. 14 days must have elapsed since discontinuation of prior chemotherapeutic treatments for glioma and study treatment.
* Radiation: Radiation is integral to the primary treatment of glioma. All participants on this study must have had prior radiation to the brain. Radiation must have been completed 14 days prior to first study treatment.
* Surgery: 14 days must have elapsed since prior major surgery.
* Organ function requirements:

  * Creatinine clearance of 50 or greater.
  * Absolute neutrophil count of 1500 or greater.
* Blood pressure requirements: Participants must have a baseline blood pressure of 160/90 or less. Participants requiring medicines to control blood pressure are eligible.
* Informed consent: All patients must sign a written informed consent.
* Urine pregnancy test: Women of childbearing age must have a negative urine pregnancy test.

Exclusion Criteria:

* People who progress with only nonenhancing tumor on MRI are ineligible. Patients must have some component of abnormal enhancement on contrast enhanced MRI of the brain. Combinations of nonenhancing and enhancing tumor are eligible.
* Pregnancy or breast-feeding: Pregnant or breast-feeding women will not be entered on this study.
* Renal insufficiency: Patients with a creatinine clearance of less than 50 are ineligible.
* Proteinuria: Patients with 2+ proteinuria/Moderate or more at baseline are ineligible.
* Comorbidities: Patients may not have any baseline comorbidities or laboratory abnormalities which would be of grade 3 or worse if graded as toxicities by CTCAE (excepting alopecia). An exception is also made for neurologic comorbidities (eg ataxia, aphasia) arising as a consequence of the brain tumor; symptoms severe enough to warrant medical treatment as is offered on this study are by definition grade 3.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Illness or any other circumstances (as defined by the investigator), which would preclude safe performance of study procedures or compromise the ability of the patient to consent to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L. Read, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institutute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at Winship Cancer Institute and Emory University Hospital Midtown from January 2014 to April 2017.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Peritumoral Enhancement/Edema
Description: To describe MRI response regarding edema and enhancement of glioblastoma and radiation-related brain enhancement when treated with subcutaneous bevacizumab daily. The therapeutic benefit of bevacizumab as regards glioblastoma multiforme (GBM) is largely due to the normalization of brain vasculature. This normalization appears on contrast-enhanced MRI as a reduction in enhancement and reduction in edema. For purposes of this study, any reduction in enhancement/edema by 25% or more will be considered a response.
Time Frame: 1 cycle (3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 3
Participants
  No change in edema | 1
  Decrease in radiation-related edema | 2

2. Secondary Outcome: Number of Toxicities Reported in Study Participants
Description: Subcutaneous bevacizumab may have toxicities unique to the subcutaneous administration and not seen with intravenous bevacizumab. During the first 3 weeks we will watch for such toxicities. Toxicities will be described and graded using the Common Toxicity Criteria for Adverse Effects (CTCAE) v3.
Time Frame: During first 3 weeks of study
Measure: Number; unit: Toxicities
Arm/Group | Bevacizumab
Number analyzed (Participants) | 3
Toxicities | 0

3. Secondary Outcome: Number of Participants With Change in Edema After Conversion From Study Treatment to Intravenous Bevacizumab
Description: Participants may switch from subcutaneous bevacizumab on study to standard of care intravenous bevacizumab. In these participants, we will measure decrease of edema after this switch. A further decrease in edema after making this switch would suggest intravenous to be superior to subcutaneous as regards decreasing edema. The therapeutic benefit of bevacizumab as regards GBM is largely due to the normalization of brain vasculature. This normalization appears on contrast-enhanced MRI as a reduction in edema. For purposes of this study, any reduction in edema by 25% or more will be considered a response.
Time Frame: Within 2 months of starting intravenous bevacizumab
Population: One patient did not switch to standard of care intravenous bevacizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 2
Participants
  No change in edema after switch | 1
  Decrease of edema after switch | 1

ADVERSE EVENTS:
Arm/Group | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=3)
Low platelets (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=3)
Bruising (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes